CLINICAL TRIAL: NCT05799365
Title: Psychometric Properties Of Turkish Adaptation Of Gross Motor Function Classification System Family Report In Children With Cerebral Palsy And The Agreement Of Family And Physiotherapist
Brief Title: Turkish Adaptation Of GMFCS Family Report And The Agreement Of Family and Physiotherapist
Status: Completed | Type: Observational
Sponsor: Muhammet Ayhan ORAL (Other)
Collaborators: Hacettepe University (Other)
Responsible Party: Sponsor-Investigator, Muhammet Ayhan ORAL, Assistant Professor, Kırıkkale University
Organization: Kırıkkale University (Other)
Other Study IDs: GMFCS-FR Turkish Adaptation
Record Dates: First submitted 2023-03-01; First posted 2023-04-05 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; Gross motor function; GMFCS; GMFCS-FR
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- 2 to 4 Years: The children with cerebral palsy between the age of 2 and 4. GMFCS-FR Turkish adaptation was applied the childrens mother, father and clinical physiotherapist.
  Interventions: Other: GMFCS-FR Turkish Adaptation
- 4 to 6 Years: The children with cerebral palsy between the age of 4 and 6. GMFCS-FR Turkish adaptation was applied the childrens mother, father and clinical physiotherapist.
  Interventions: Other: GMFCS-FR Turkish Adaptation
- 6 to 12 Years: The children with cerebral palsy between the age of 6 and 12. GMFCS-FR Turkish adaptation was applied the childrens mother, father and clinical physiotherapist.
  Interventions: Other: GMFCS-FR Turkish Adaptation
- 12 to 18 Years: The children with cerebral palsy between the age of 12 and 18. GMFCS-FR Turkish adaptation was applied the childrens mother, father and clinical physiotherapist.
  Interventions: Other: GMFCS-FR Turkish Adaptation
- 12 to 18 Years Young with Good Cognitive Levels: The children with cerebral palsy with good cognitive levels between the age of 12 and 18. GMFCS-FR Turkish adaptation was applied the childrens mother, father and clinical physiotherapist.
  Interventions: Other: GMFCS-FR Turkish Adaptation

INTERVENTIONS:
Other: GMFCS-FR Turkish Adaptation — GMFCS-FR Turkish Adaptation was applied the childrens mother, father and clinical physiotherapist.

SUMMARY:
To make the Turkish adaptation of the Gross Motor Function Classification System Family Report (GMFCS-FR) in children with CP, to determine its reliability and validity, and to investigate the agreement of the family and the clinical physiotherapists in determining the gross motor function level.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a heterogeneous, persistent neurological disorder caused by non-progressive damage to the developing brain. This condition occurs as a result of injury or malformation in the developing central nervous system before, during or immediately after birth. This situation, which develops secondary to lesions or abnormalities of the central nervous system, affects motor function and posture development. As a result of the addition of tertiary disorders to the table with different compensation mechanisms over time, the development and functional independence levels of children are negatively affected.

Diagnosis in CP can be made in the first two years of life, especially when functional impairment is mild. However, there is a consensus that 5 years of age is the most appropriate age to confirm the diagnosis, due to the clinical condition that may change with the development of the child in some cases.

Since recent studies on the rehabilitation of children with CP have focused on increasing functionality in their daily activities, the functional levels and abilities of these children have recently gained more importance. It may be necessary to use some test batteries in order to evaluate the motor development and functional level of the child. Gross Motor Function Classification System (GMFCS) used for functional classification and Pediatric Functional Independence Measure (WeeFIM) used for pediatric functional evaluation of activities of daily living are some of the commonly used test batteries.

In the last 20 years, family-centered approaches have gained importance for children with CP and their families. Family-centered approaches that address the needs of children and their families, and families' involvement in all aspects of services for their children contribute to the establishment of partnership between parents and health professionals. Family-assessed measurements or family reports are invaluable, as families are at the center of the rehabilitation process, with active participation in all phases of CP treatment and management. Therefore, it becomes important to investigate the validity, reliability and stability of classification systems that can also be used by parents.

GMFCS, which is widely used in research and clinical practice for treatment and rehabilitation planning, prognosis and clinical decision making, was modified in 2004 by Morris et al. to be used for parents and named GMFCS Family Report Questionnaire.

The aim of this study is to make the Turkish adaptation of the Gross Motor Function Classification System Family Report (GMFCS-FR) in children with CP, to determine its reliability and validity, and to investigate the agreement of the family and the clinical physiotherapists in determining the gross motor function level.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with cerebral palsy between the ages of 2 and 18 who agreed to participate in the study
* Clinical physiotherapists of of children with cerebral palsy between the ages of 2 and 18 who agreed to participate in the study

Exclusion Criteria:

* refuse to participate in the study
* Parents of individuals with cerebral palsy who are not between the ages of 2 and 18

Ages: 2 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: The study was terminated with the participation of a total of 100 children's parents (mother and father), 18 clinical physiotherapists and 20 young people with CP between the ages of 12 to 18 years with good cognitive level.
  Children with CP were divided into four different age groups. 2 to 4 years of age, 4 to 6 years of age, 6 to 12 years of age and 12 to 18 years of age were determined and all examinations were performed according to these groups. A fifth group of GMFCS-FR created for young people aged 12 to 18 years with good cognitive level is called GMFCS-FR self-report. The young people aged 12 to 18 in our study with good cognitive level were included in the 5th group. Each group consisted of 20 children with CP
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Change in GMFCS-FR Turkish Adaptation Reliability | 30 minutes
  For test-retest reliability, the mothers and fathers of each of the 100 children with CP who participated in the study, and young people aged 12 to 18 years with good cognitive level were asked to answer the GMFCS-FR twice, with an interval of 15 days.

SECONDARY OUTCOMES:
GMFCS-FR Turkish Adaptation Inter-Observer Reliability | 30 minutes
  ICC values were used to determine the interobserver reliability of the questionnaire. The GMFCS levels recorded by the research physiotherapist by learning from the children's clinical physiotherapists and the GMFCS-FR levels determined by mothers, fathers and young people aged 12 to 18 years with good cognitive level were compared.

OTHER OUTCOMES:
GMFCS-FR Turkish Adaptation Validity | 30 minutes
  The concurrent validity of the GMFCS-FR was evaluated with the Pediatric Functional Independence Measure (WeeFIM 2®). WeeFIM 2® scores were compared with the GMFCS-FR levels determined separately by each of the mothers, fathers and 12 to 18 Years Young with Good Cognitive Levels GMFCS FR-SR. Spearman's Correlation Coefficient was used for analysis.
Agreement of GMFCS-FR Levels Determined by Mothers, Fathers, young people aged 12 to 18 years with good cognitive level and Clinical physiotherapist | 30 minutes
  Kappa values were calculated for agreement between GMFCS-FR levels determined individually by each participant
The Relationship between the GMFCS-FR Levels Determined by Clinical Physiotherapists and the GMFCS Levels Determined by Clinical Physiotherapists | 30 minutes
  When the relationship between the GMFCS-FR levels of the child determined by the clinical physiotherapists participating in the study and the GMFCS levels was examined

CONTACTS AND LOCATIONS:
Overall Officials: MINTAZE KEREM GUNEL, PROF, Study Director — Hacettepe University
Locations (1):
- Hacettepe University Faculty of Physical Therapy and Rehabilitaton, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Alriksson-Schmidt A, Nordmark E, Czuba T, Westbom L. Stability of the Gross Motor Function Classification System in children and adolescents with cerebral palsy: a retrospective cohort registry study. Dev Med Child Neurol. 2017 Jun;59(6):641-646. doi: 10.1111/dmcn.13385. Epub 2017 Jan 13. PMID 28083887
- [Background] Livanelioğlu A, Fizyoterapi KGMSP. Ankara. Yeni Özbek Matbaası
- [Background] Ford GW, Kitchen WH, Doyle LW, Rickards AL, Kelly E. Changing diagnosis of cerebral palsy in very low birthweight children. Am J Perinatol. 1990 Apr;7(2):178-81. doi: 10.1055/s-2007-999475. PMID 2331281
- [Background] Jacobsson B, Hagberg G. Antenatal risk factors for cerebral palsy. Best Pract Res Clin Obstet Gynaecol. 2004 Jun;18(3):425-36. doi: 10.1016/j.bpobgyn.2004.02.011. PMID 15183137
- [Background] Christine C, Dolk H, Platt MJ, Colver A, Prasauskiene A, Krageloh-Mann I; SCPE Collaborative Group. Recommendations from the SCPE collaborative group for defining and classifying cerebral palsy. Dev Med Child Neurol Suppl. 2007 Feb;109:35-8. doi: 10.1111/j.1469-8749.2007.tb12626.x. No abstract available. PMID 17370480
- [Background] Mayston MJ. People with cerebral palsy: effects of and perspectives for therapy. Neural Plast. 2001;8(1-2):51-69. doi: 10.1155/NP.2001.51. PMID 11530888
- [Background] Mayston MJ. Bobath Concept Theory Clinical Practice in Neurological Rehabilitation: Synapse, Spring; 2001. 32-4 p.
- [Background] Ottenbacher KJ, Msall ME, Lyon NR, Duffy LC, Granger CV, Braun S. Interrater agreement and stability of the Functional Independence Measure for Children (WeeFIM): use in children with developmental disabilities. Arch Phys Med Rehabil. 1997 Dec;78(12):1309-15. doi: 10.1016/s0003-9993(97)90302-6. PMID 9421983
- [Background] King G, Chiarello L. Family-centered care for children with cerebral palsy: conceptual and practical considerations to advance care and practice. J Child Neurol. 2014 Aug;29(8):1046-54. doi: 10.1177/0883073814533009. Epub 2014 May 7. PMID 24810084
- [Background] Rosenbaum P, King S, Law M, King G, Evans J. Family-centred service: A conceptual framework and research review. Physical & Occupational Therapy in Pediatrics. 1998;18(1):1-20.
- [Background] Mutlu A, Kara OK, Gunel MK, Karahan S, Livanelioglu A. Agreement between parents and clinicians for the motor functional classification systems of children with cerebral palsy. Disabil Rehabil. 2011;33(11):927-32. doi: 10.3109/09638288.2010.514645. Epub 2010 Sep 3. PMID 20815692
- [Background] Wiart L, Ray L, Darrah J, Magill-Evans J. Parents' perspectives on occupational therapy and physical therapy goals for children with cerebral palsy. Disabil Rehabil. 2010;32(3):248-58. doi: 10.3109/09638280903095890. PMID 20001831
- [Background] Morris C, Bartlett D. Gross Motor Function Classification System: impact and utility. Dev Med Child Neurol. 2004 Jan;46(1):60-5. doi: 10.1017/s0012162204000118. PMID 14974650
- [Background] Morris C, Galuppi BE, Rosenbaum PL. Reliability of family report for the Gross Motor Function Classification System. Dev Med Child Neurol. 2004 Jul;46(7):455-60. doi: 10.1017/s0012162204000751. PMID 15230458
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Palisano RJ, Cameron D, Rosenbaum PL, Walter SD, Russell D. Stability of the gross motor function classification system. Dev Med Child Neurol. 2006 Jun;48(6):424-8. doi: 10.1017/S0012162206000934. PMID 16700931
- [Background] Palisano RJ, Rosenbaum P, Bartlett D, Livingston MH. Content validity of the expanded and revised Gross Motor Function Classification System. Dev Med Child Neurol. 2008 Oct;50(10):744-50. doi: 10.1111/j.1469-8749.2008.03089.x. PMID 18834387
- [Background] Akpinar P, Tezel CG, Eliasson AC, Icagasioglu A. Reliability and cross-cultural validation of the Turkish version of Manual Ability Classification System (MACS) for children with cerebral palsy. Disabil Rehabil. 2010;32(23):1910-6. doi: 10.3109/09638281003763796. PMID 20373857
- [Background] Wong V, Wong S, Chan K, Wong W. Functional Independence Measure (WeeFIM) for Chinese children: Hong Kong Cohort. Pediatrics. 2002 Feb;109(2):E36. doi: 10.1542/peds.109.2.e36. PMID 11826246
- [Background] Lin HY, Lin SP, Lin HY, Hsu CH, Chang JH, Kao HA, Hung HY, Peng CC, Lee HC, Chen MR, Tsai JD. Functional independence of Taiwanese children with VACTERL association. Am J Med Genet A. 2012 Dec;158A(12):3101-5. doi: 10.1002/ajmg.a.33643. Epub 2012 Nov 19. PMID 23165933
- [Background] Ottenbacher KJ, Msall ME, Lyon N, Duffy LC, Granger CV, Braun S. Measuring developmental and functional status in children with disabilities. Dev Med Child Neurol. 1999 Mar;41(3):186-94. doi: 10.1017/s0012162299000377. PMID 10210251
- [Background] Morris C, Kurinczuk JJ, Fitzpatrick R, Rosenbaum PL. Who best to make the assessment? Professionals' and families' classifications of gross motor function in cerebral palsy are highly consistent. Arch Dis Child. 2006 Aug;91(8):675-9. doi: 10.1136/adc.2005.090597. Epub 2006 Apr 25. PMID 16638783
- [Background] Ramrit S, Yonglitthipagon P, Janyacharoen T, Emasithi A, Siritaratiwat W. The Gross Motor Function Classification System Family Report Questionnaire: reliability between special-education teachers and caregivers. Dev Med Child Neurol. 2017 May;59(5):520-525. doi: 10.1111/dmcn.13356. Epub 2016 Dec 14. PMID 27966216
- [Background] Oksuz C, Alemdaroglu I, Kilinc M, Abaoglu H, Demirci C, Karahan S, Yilmaz O, Yildirim SA. Reliability and validity of the Turkish version of ABILHAND-Kids' questionnaire in a group of patients with neuromuscular disorders. Physiother Theory Pract. 2017 Oct;33(10):780-787. doi: 10.1080/09593985.2017.1346026. Epub 2017 Jul 17. PMID 28715270
- [Background] Gunel MK, Mutlu A, Tarsuslu T, Livanelioglu A. Relationship among the Manual Ability Classification System (MACS), the Gross Motor Function Classification System (GMFCS), and the functional status (WeeFIM) in children with spastic cerebral palsy. Eur J Pediatr. 2009 Apr;168(4):477-85. doi: 10.1007/s00431-008-0775-1. Epub 2008 Jun 13. PMID 18551314